CLINICAL TRIAL: NCT01294384
Title: Safety and Efficacy Study of New Eye Drop Formulations With Refresh Tears® in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10078X-001
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- New Eye Drop Formulation 1 (Experimental): 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation 1 in each eye at least twice daily for 90 days.
  Interventions: Drug: carboxymethylcellulose sodium based New Eye Drop Formulation 1
- New Eye Drop Formulation 2 (Experimental): 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation 2 in each eye at least twice daily for 90 days.
  Interventions: Drug: carboxymethylcellulose sodium based New Eye Drop Formulation 2
- Refresh Tears® (Active Comparator): 1 to 2 drops of carboxymethylcellulose sodium based Eye Drops (Refresh Tears®) in each eye at least twice daily for 90 days.
  Interventions: Drug: carboxymethylcellulose sodium based Eye Drops

INTERVENTIONS:
Drug: carboxymethylcellulose sodium based New Eye Drop Formulation 1 — 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation 1 in each eye at least twice daily for 90 days.
  Arms: New Eye Drop Formulation 1
Drug: carboxymethylcellulose sodium based New Eye Drop Formulation 2 — 1 to 2 drops of carboxymethylcellulose sodium based New Eye Drop Formulation 2 in each eye at least twice daily for 90 days.
  Arms: New Eye Drop Formulation 2
Drug: carboxymethylcellulose sodium based Eye Drops — 1 to 2 drops of carboxymethylcellulose sodium based Eye Drops (Refresh Tears®) in each eye at least twice daily for 90 days.
  Other Names: Refresh Tears®
  Arms: Refresh Tears®

SUMMARY:
This study will investigate the safety, efficacy and acceptability of two new eye drop formulations compared with Refresh Tears® in patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Current use of an artificial tear product at least twice daily for at least 3 months, on average
* Ability/agreement to continue wearing existing spectacle correction (glasses) during study

Exclusion Criteria:

* Anticipated contact lens wear during study or contact lens use within 6 months
* Active ocular infection or allergy
* Use of any topical ophthalmic medications (eg, topical ophthalmic steroids, glaucoma drops) within 2 weeks
* Use of any topical cyclosporine products within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2012-09-25 (Actual); Study Completion 2012-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (2):
- Randwick, New South Wales, Australia
- St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Background] Simmons PA, Liu H, Carlisle-Wilcox C, Vehige JG. Efficacy and safety of two new formulations of artificial tears in subjects with dry eye disease: a 3-month, multicenter, active-controlled, randomized trial. Clin Ophthalmol. 2015 Apr 15;9:665-75. doi: 10.2147/OPTH.S78184. eCollection 2015. PMID 25931807

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Started | 101 | 100 | 104
Completed | 97 | 94 | 95
Not Completed | 4 | 6 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears® | Total
Number analyzed (Participants) | 101 | 100 | 104 | 305
Age, Customized [Number; unit: Participants]
  < 40 years | 9 | 13 | 7 | 29
  40 to 60 years | 42 | 33 | 43 | 118
  > 60 years | 50 | 54 | 54 | 158
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 80 | 90 | 248
  Male | 23 | 20 | 14 | 57

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Ocular Surface Disease Index© (OSDI) Score
Description: The OSDI is a questionnaire consisting of 12 questions assessing severity of dry eye using a 5-point scale where 0=none of the time to 4=all of the time. The total score is the sum of the individual scores normalized (standardized) to a severity scale of 0=no symptoms (best score) to 100=maximum severity (worst score). A negative change from Baseline indicated improvement.
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Score on a scale
  Baseline | 36.83 (13.350) | 38.51 (12.512) | 38.86 (11.880)
  Change from Baseline at Day 90 | -14.72 (16.319) | -12.75 (17.612) | -14.49 (16.443)

2. Secondary Outcome: Change From Baseline in Visual Analog (VAS) Symptom Scale: Dryness
Description: The participant rated the severity of their dry eye symptom: dryness using a VAS scale. Participants put a mark on a 100 millimeter line where 0 (far left on the line)=no symptoms to 100 (far right on the line)=most severe symptoms.
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
millimeters
  Baseline | 61.1 (22.10) | 64.0 (19.05) | 60.9 (18.98)
  Change from Baseline at Day 90 | -24.2 (30.78) | -19.2 (29.44) | -20.9 (29.20)

3. Secondary Outcome: Percentage of Participants Much Better or Better in Near Visual Acuity (Low Contrast)
Description: Near Visual Acuity was determined using the number of letters read correctly on a low contrast eye chart (gray letters on a white background). An increase in the number of letters read correctly indicated improvement. Much Better is defined as an increase of 10 or more letters read correctly at Day 90 compared to the worse eye at Baseline. Better is defined as an increase of 5 to 9 letters read correctly at Day 90 compared to the worse eye at Baseline.
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Percentage of participants
  Much better | 5.0 | 8.0 | 5.8
  Better | 22.0 | 21.0 | 30.8

4. Secondary Outcome: Percentage of Participants Much Better or Better in Near Visual Acuity (High Contrast)
Description: Near Visual Acuity was determined using the number of letters read correctly on a high contrast eye chart (black letters on a white background). An increase in the number of letters read correctly indicated improvement. Much Better is defined as an increase of 10 or more letters read correctly at Day 90 compared to the worse eye at Baseline. Better is defined as an increase of 5 to 9 letters read correctly at Day 90 compared to the worse eye at Baseline.
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Percentage of participants
  Much Better | 7.0 | 6.0 | 4.8
  Better | 15.0 | 20.0 | 22.1

5. Secondary Outcome: Change From Baseline in Tear Break-Up Time (TBUT)
Description: TBUT is defined as the time (seconds) required for dry spots to appear on the surface of the eye after blinking. The longer it takes, the more stable the tear film. A positive number change from Baseline indicated improvement.
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Seconds
  Baseline | 5.24 (2.007) | 5.22 (1.870) | 5.05 (1.894)
  Change from Baseline at Day 90 | 1.65 (4.268) | 1.97 (3.294) | 1.27 (2.837)

6. Secondary Outcome: Change From Baseline in Corneal Staining
Description: The cornea is the transparent front part of the eye which covers the iris and pupil. Corneal staining following administration of fluorescein dye in the eye is graded using a 6-point scale where 0=no staining to 5=severe staining over 5 areas of the clear central part of the eye for a minimum score of 0 and maximum score of 25. The higher the grade score, the worse the dry eye condition. A negative number change from baseline represented a decrease in corneal staining (improvement).
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Score on a scale
  Baseline | 6.4 (4.97) | 6.1 (4.25) | 5.8 (4.29)
  Change from Baseline at Day 90 | -2.3 (3.75) | -2.0 (3.36) | -1.2 (3.13)

7. Secondary Outcome: Change From Baseline in Conjunctival Staining
Description: The conjunctiva is the clear membrane covering the white surface of the eye. Conjunctival staining following ocular administration of lissamine green dye was graded using a 6-point scale where 0=no staining to 5=severe staining over 6 areas of the white part of the eye for a minimum score of 0 and a maximum score of 30. The higher the score, the worse the dry eye condition. A negative number change from baseline represented a decrease in the severity of conjunctival staining (improvement).
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
Score on a scale
  Baseline | 8.0 (5.34) | 7.8 (5.45) | 8.2 (5.44)
  Change from Baseline at Day 90 | -2.7 (4.72) | -2.4 (4.06) | -2.7 (4.36)

8. Secondary Outcome: Change From Baseline in Schirmer Test
Description: The Schirmer Test measures the rate of the secretion of tears produced by the eye over 5 minutes. The results indicate the presence of dry eye where Normal=greater than or equal to 10 millimeters (mm) of tears and Dry Eye=less than 10 mm of tears). The smaller the number, the more severe the dry eye. A positive number change from baseline indicated an increase in tears (improvement).
Time Frame: Baseline, Day 90
Population: Participants from the Intent-to-Treat population, that included all randomized participants.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Number analyzed (Participants) | 101 | 100 | 104
mm
  Baseline | 8.7 (6.96) | 10.3 (7.17) | 8.9 (6.16)
  Change from Baseline at Day 90 | 1.2 (7.07) | 1.5 (6.12) | 1.1 (7.07)

ADVERSE EVENTS:
Description: The safety population, that included all participants who received at least one dose of study treatment, was used to calculate the number of participants at risk for Adverse Events. (One randomized patient did not receive treatment and two patients received treatment but were not randomized.)
Arm/Group | New Eye Drop Formulation 1 | New Eye Drop Formulation 2 | Refresh Tears®
Serious Adverse Events (participants affected / at risk) | 2/102 | 2/101 | 1/103
Other Adverse Events (participants affected / at risk) | 0/102 | 0/101 | 0/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Eye Drop Formulation 1 (N=102) | New Eye Drop Formulation 2 (N=101) | Refresh Tears® (N=103)
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.